CLINICAL TRIAL: NCT06336577
Title: Infectious and Non-infectious Lower Respiratory Diseases in Children With Down Syndrome Followed in Pediatric Pulmonology Consultations in Ile-de-France
Acronym: ARBT21
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0003
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Down Syndrome
Keywords: Down syndrome; children; lower respiratory diseases; respiratory infection; respiratory syncytial virus; hemosiderosis; asthma; bronchiolitis
MeSH Terms: conditions — Down Syndrome; Respiratory Tract Infections; Hemosiderosis; Asthma; Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lower respiratory tract disease — lower respiratory tract disease

SUMMARY:
The purpose of this study is to describe infectious and non-infectious lower respiratory tract diseases in children with Down syndrome followed in pediatric pulmonology consultations in Ile de France.

DETAILED DESCRIPTION:
Down syndrome is the most common chromosomal abnormality, affecting 600 to 800 births per year. It results in a clinical picture that combines developmental delay, mental deficiency, facial dysmorphism and visceral malformations.

Optimal medical care of Down syndrome patients requires a good knowledge of the different systems affected by the disease, particularly respiratory damage.

Numerous articles have been published describing upper respiratory problems in children with Down syndrome. On the other hand, lower respiratory problems causing significant morbidity and mortality remain underestimated and poorly understood in this population.

The objective of this study is to describe lower respiratory problems in patients with T21, in order to improve their management.

This study will also make it possible to describe more precisely the impact that these attacks have on Down syndrome patients.

This study also describe the associated extra-respiratory disorders to improve overall care Finally, the respiratory care of these patients will be described, with the aim of standardizing practices.

ELIGIBILITY:
Inclusion Criteria:

* Child from 0 to 17 years old
* Carrier of Down syndrome confirmed by karyotype
* Having had follow-up in a pediatric pulmonology consultation for an infectious or non-infectious lower respiratory tract
* Not exclusively presenting upper respiratory otorhinolaryngological damage

Exclusion Criteria:

* Patient under guardianship or curators
* Adult or holders of parental authority informed of the study and having objected to it

Ages: 1 Day to 17 Years | Sex: All
Age Groups: Child
Study Population: children with Down syndrome, who were hospitalized for respiratory problems and who had subsequent pediatric pulmonology follow-up between 2013 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
distribution of lower respiratory tract diseases | at day 0
  number

CONTACTS AND LOCATIONS:
Overall Officials: Yousra MESBAHI, MD, Principal Investigator — C
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No